CLINICAL TRIAL: NCT06134128
Title: Compensatory Cognitive Training Via Telehealth for Veterans With Alcohol Use Disorders (CCT-A)
Brief Title: Compensatory Cognitive Training Via Telehealth for Veterans With Alcohol Use Disorders
Acronym: CCT-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kate Shirley, Principal Investigator, Portland VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6208
Record Dates: First submitted 2023-09-18; First posted 2023-11-18 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder
Keywords: cognitive rehabilitation
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motivationally Enhanced Compensatory Cognitive Training for Addictions Group (Experimental): Motivationally Enhanced Compensatory Cognitive Training for Addictions (ME-CCT-A) is a manualized group-based behavioral intervention (8 weeks, 2 hour per week) designed to improve cognitive functioning in Veterans with substance use disorders (SUDs) and cognitive complaints.
  Interventions: Behavioral: Motivationally Enhanced Compensatory Cognitive Training for Addictions Group

INTERVENTIONS:
Behavioral: Motivationally Enhanced Compensatory Cognitive Training for Addictions Group — 8-week manualized group-based behavioral intervention delivered via telehealth

SUMMARY:
Most individuals entering treatment for alcohol use disorders (AUDs) present with cognitive deficits across a range of cognitive domains, and these deficits frequently persist for six months or longer following remission. Cognitive deficits are associated with increased relapse rates, less treatment compliance, and poorer treatment outcomes in individuals seeking substance use treatment. Despite the high rates of cognitive impairments among adults with AUDs and their negative impact on treatment outcomes, current evidence-based treatments for AUDs do not specifically treat or address cognitive symptoms. Accessible (e.g., brief, manualized, delivered via telehealth) and effective treatments for adults with AUDs and cognitive deficits are urgently needed.

The primary objective of this study is to assess the feasibility and acceptability of a manualized, 8-week, Compensatory Cognitive Training (CCT) intervention delivered via telehealth for Veterans in early remission from alcohol use disorder (AUD).

The investigators hypothesize that Motivationally Enhanced Compensatory Cognitive Training for Addictions (ME-CCT-A) will be feasible and acceptable in a pilot trial of ME-CCT-A delivered via telehealth.

DETAILED DESCRIPTION:
Motivationally Enhanced Compensatory Cognitive Training for Addictions (ME-CCT-A) is a manualized group-based behavioral intervention (8 weeks, 2 hour per week) designed to improve cognitive functioning in Veterans with substance use disorders (SUDs) and cognitive complaints. ME-CCT-A is an adaptation of CCT initially developed by clinicians and researchers at the VA Portland Healthcare System and VA San Diego Healthcare System. CCT draws from the empirical and theoretical literature on compensatory strategy training for conditions characterized by cognitive complaints and impairments, including mild traumatic brain injury, psychosis, and mild cognitive impairment. ME-CCT-A is a comprehensive treatment in that it addresses multiple types of symptoms and concerns that interfere with recovery from addictions - cognitive impairments, neuropsychiatric symptoms, and lifestyle patterns that increase risk of cognitive impairment, poor health, and relapse. In addition to training in compensatory cognitive skills, ME-CCT-A includes mindfulness practices and motivational interviewing techniques to boost the adoption of lifestyle strategies (e.g., nutrition, exercise) that improve cognition and overall health. ME-CCT-A is designed to be easy to administer and as an adjunct to standard SUD treatment programs. While initially designed to be delivered in-person, ME-CCT-A can be delivered through virtual platforms with little to no modification of the content and structure of the intervention.

Given the high rate of AUDs among Veterans, the prevalence of cognitive impairments among those with AUDs, and the negative impact of cognitive impairments on treatment outcomes, an evidence-based cognitive training intervention that optimally addresses the complex needs of Veterans with AUDs and cognitive impairments is of critical importance. This study will allow the investigators to optimize ME-CCT-A for the telehealth format and assess the feasibility and acceptability of the intervention in preparation for a larger-scale pilot randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Veterans (>18 years) who meet criteria for AUD in early remission (>1 month, <12 months remission) based on the DSM-5 (American Psychiatric Association, 2013)
* Concern about a mild cognitive decline that has been identified by the Veteran or a knowledgeable informant (e.g., SUD treatment providers), and the Veteran wants treatment for their cognitive concerns
* Access to internet and webcam.

Exclusion Criteria:

* Intoxication or impaired capacity to understand study risks and benefits
* Major Neurocognitive Disorder, dementia, neurodegenerative disorder (e.g., Alzheimer's Disease)
* Auditory or visual impairments that would prevent ability to participate in the cognitive rehabilitation group or benefit from compensatory strategies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Portland VA Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Motivationally Enhanced Compensatory Cognitive Training for Addictions Group
Started | 19
Completed | 15
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Motivationally Enhanced Compensatory Cognitive Training for Addictions Group
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Education [Mean (Standard Deviation); unit: years] — Years of education
  years | 13.9 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: Number of participants included from eligible Veterans; satisfactory recruitment defined as enrolment of ≥ 50% of eligible Veterans.
Time Frame: From enrollment to the end of treatment at 8 weeks
Population: Thirty-two individuals expressed interest, and 29 completed screening; 19 Veterans enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivationally Enhanced Compensatory Cognitive Training for Addictions Group
Number analyzed (Participants) | 29
Participants | 19

2. Primary Outcome: Study Retention
Description: Satisfactory retention rate ≥ 75% of participants completing the intervention.
Time Frame: From enrollment to the end of treatment at 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Motivationally Enhanced Compensatory Cognitive Training for Addictions Group
Number analyzed (Participants) | 19
Participants | 15

3. Primary Outcome: Feasibility of Testing Procedures
Description: % of participants where follow-up visit was completed.
Time Frame: From enrollment to the end of treatment at 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Motivationally Enhanced Compensatory Cognitive Training for Addictions Group
Number analyzed (Participants) | 19
Participants | 15

4. Primary Outcome: Feasibility of Data Collection Methods
Description: % of participants with complete data sets.
Time Frame: From enrollment to the end of treatment at 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Motivationally Enhanced Compensatory Cognitive Training for Addictions Group
Number analyzed (Participants) | 19
Participants | 15

5. Primary Outcome: Acceptability, by Participant Report
Description: Satisfactory acceptability ≥ 70% of participants score ≥ 24 on the Client Satisfaction Questionnaire (CSQ-8). CSQ-8 scores range from 8-32, with higher scores indicating greater satisfaction with the intervention.
Time Frame: Measured after the 8-week intervention
Measure: Number; unit: participants' score ≥ 24
Arm/Group | Motivationally Enhanced Compensatory Cognitive Training for Addictions Group
Number analyzed (Participants) | 15
participants' score ≥ 24 | 15

ADVERSE EVENTS:
Time Frame: 1 year
Description: All adverse events were reported immediately to the Co-PIs who evaluated the patient and determined if any additional evaluation or treatment was needed. Co-PIs ensured that adverse events were properly reported to the IRB. The study staff examined all cumulative adverse events quarterly to determine if there were any systematic problems.
Arm/Group | Motivationally Enhanced Compensatory Cognitive Training for Addictions Group
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

LIMITATIONS AND CAVEATS:
The small sample size reduced statistical power and generalizability, although this is consistent with early stage feasibility research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT06134128/Prot_SAP_000.pdf